CLINICAL TRIAL: NCT02990780
Title: Phase III Randomized Study of Induction Chemotherapy Followed By Accelerated Hypofractionated vs. Conventionally Fractionated Concurrent Chemo-radiotherapy for Limited Stage Small Cell Lung Cancer.
Brief Title: Accelerated Hypofractionated vs. Conventionally Fractionated Concurrent CRT for LS-SCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Fu, Director, Department of Radiation Oncology, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHLC010
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: SCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventionally fractionated CRT (Active Comparator): Induction chemotherapy followed by conventionally fractionated concurrent chemo-radiotherapy,with prophylactic cranial irradiation for those who achieve a good response after combined chemoradiotherapy.
  Interventions: Radiation: Conventionally fractionated concurrent chemo-radiotherapy
- Accelerated hypofractionated CRT (Experimental): Induction chemotherapy followed by accelerated hypofractionated concurrent chemo-radiotherapy,with prophylactic cranial irradiation for those who achieve a good response after combined chemoradiotherapy.
  Interventions: Radiation: Accelerated hypofractionated concurrent chemo-radiotherapy

INTERVENTIONS:
Radiation: Conventionally fractionated concurrent chemo-radiotherapy — 5Fx/W,2Gy/Fx,Dt:PTV-G:60Gy/30F/6W.
  Arms: Conventionally fractionated CRT
Radiation: Accelerated hypofractionated concurrent chemo-radiotherapy — 5Fx/W,2.5Gy/Fx,Dt:PTV-G:55Gy/22F/4.4W.
  Arms: Accelerated hypofractionated CRT

SUMMARY:
This protocol is a phase III randomized controlled trial (RCT) evaluating the efficacy of induction chemotherapy followed by accelerated hypofractionated vs. conventionally fractionated concurrent chemo-radiotherapy for limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
Small-cell lung cancer accounts for approximately 13% of all lung cancers, and one-third of these patients present with limited stage SCLC at diagnosis. Currently the standard of care for LS-SCLC is concurrent chemotherapy and thoracic radiation therapy, with prophylactic cranial irradiation for those who achieve a good response after combined chemoradiotherapy, which has yielded a median survival of 15 to 23 months and 5-year survival rate up to 26%.

The optimal dose/fraction for LS-SCLC remains debatable. For SCLC with the characteristic of rapid doubling time and high growth fraction, there is also evidence suggesting that prolonged or interrupted overall radiation time contributes to treatment failure and poor outcome because of accelerated repopulation.In our previous study we also found that overall radiation time might play an important role in the treatment of LS-SCLC and that patients treated with a high biologically effective dose (BED, including time factor) of >57 Gy have favorable local control and survival.

This is a randomised prospective phase III study based on patients with limited stage SCLC, defined as disease confined to one hemithorax and hilar,mediastinal, or supraclavicular nodes without pleural effusion, which can be safely encompassed within a tolerable radiation field. The purpose of this study is to add more information to the current medical literature about the efficacy and safety of accelerated hypofractionated vs. conventionally fractionated concurrent chemo-radiotherapy for limited-stage SCLC.

Patients will be randomized into two groups. The control group will undergo the induction chemotherapy followed by conventionally fractionated concurrent chemo-radiotherapy.The experimental group will receive induction chemotherapy followed by accelerated hypofractionated concurrent chemo-radiotherapy.The investigators compare overall survival (OS) of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed SCLC.
* Male or female, aged 18-70 years.
* ECOG performance status 0 to 2.
* Limited-stage SCLC was defined as disease confined to one hemithorax and hilar,mediastinal, or supraclavicular nodes without pleural effusion, which can be safely encompassed within a tolerable radiation field.
* No prior thoracic RT.
* Weight loss in six months less than or equal to five percent.
* FEV1 greater than 0.75L.
* No severe internal diseases and no organ dysfunction.
* No prior history of any tumor.
* Skin test of CT contrast agents was negative.
* Had received 1-6 cycles of VP16 plus DDP/carboplatin.
* Voluntarily participated in this study and signed the informed consent form by himself or his agent. Had good compliance with the study procedures, and can cooperate with the relevant examination, treatment and follow-up.

Exclusion Criteria:

* Other tumor history(Except skin cancer/breast cancer/oral cancer/cervical cancer with expected lifespan more than or equal to 3 months).
* Multiple primary lung cancer.
* Any unstable systemic disease, including active infection, uncontrolled high blood pressure, unstable angina, newly observed angina pectoris within the past 3 months, congestive heart failure (New York heart association (NYHA) class II or higher), myocardial infarction onset six months before included into the group, and severe arrhythmia, liver, kidney, or metabolic disease in need of drug therapy. Human immunodeficiency virus (HIV) infection.
* Women in pregnancy or lactation .
* Patients with mental illness, considered as "can't fully understand the issues of this research".
* Had received other chemotherapy regimens,any radiotherapy or TKI.
* Refuse to write informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years

SECONDARY OUTCOMES:
Progress Free Survival | 2 years
Treatment-related adverse event | 1 years
Locoregional recurrence-free survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Govindan R, Page N, Morgensztern D, Read W, Tierney R, Vlahiotis A, Spitznagel EL, Piccirillo J. Changing epidemiology of small-cell lung cancer in the United States over the last 30 years: analysis of the surveillance, epidemiologic, and end results database. J Clin Oncol. 2006 Oct 1;24(28):4539-44. doi: 10.1200/JCO.2005.04.4859. PMID 17008692
- [Background] Bayman NA, Sheikh H, Kularatne B, Lorigan P, Blackhall F, Thatcher N, Faivre-Finn C. Radiotherapy for small-cell lung cancer-Where are we heading? Lung Cancer. 2009 Mar;63(3):307-14. doi: 10.1016/j.lungcan.2008.06.013. Epub 2008 Aug 3. PMID 18676057
- [Background] Stinchcombe TE, Gore EM. Limited-stage small cell lung cancer: current chemoradiotherapy treatment paradigms. Oncologist. 2010;15(2):187-95. doi: 10.1634/theoncologist.2009-0298. Epub 2010 Feb 9. PMID 20145192
- [Background] Mamdani H, Induru R, Jalal SI. Novel therapies in small cell lung cancer. Transl Lung Cancer Res. 2015 Oct;4(5):533-44. doi: 10.3978/j.issn.2218-6751.2015.07.20. PMID 26629422
- [Background] Semenova EA, Nagel R, Berns A. Origins, genetic landscape, and emerging therapies of small cell lung cancer. Genes Dev. 2015 Jul 15;29(14):1447-62. doi: 10.1101/gad.263145.115. PMID 26220992
- [Background] Pietanza MC, Byers LA, Minna JD, Rudin CM. Small cell lung cancer: will recent progress lead to improved outcomes? Clin Cancer Res. 2015 May 15;21(10):2244-55. doi: 10.1158/1078-0432.CCR-14-2958. PMID 25979931
- [Background] Kalemkerian GP. Advances in pharmacotherapy of small cell lung cancer. Expert Opin Pharmacother. 2014 Nov;15(16):2385-96. doi: 10.1517/14656566.2014.957180. Epub 2014 Sep 26. PMID 25255939
- [Background] Pignon JP, Arriagada R, Ihde DC, Johnson DH, Perry MC, Souhami RL, Brodin O, Joss RA, Kies MS, Lebeau B, et al. A meta-analysis of thoracic radiotherapy for small-cell lung cancer. N Engl J Med. 1992 Dec 3;327(23):1618-24. doi: 10.1056/NEJM199212033272302. PMID 1331787
- [Background] Warde P, Payne D. Does thoracic irradiation improve survival and local control in limited-stage small-cell carcinoma of the lung? A meta-analysis. J Clin Oncol. 1992 Jun;10(6):890-5. doi: 10.1200/JCO.1992.10.6.890. PMID 1316951
- [Background] Xia B, Chen GY, Cai XW, Zhao JD, Yang HJ, Fan M, Zhao KL, Fu XL. The effect of bioequivalent radiation dose on survival of patients with limited-stage small-cell lung cancer. Radiat Oncol. 2011 May 19;6:50. doi: 10.1186/1748-717X-6-50. PMID 21592406
- [Background] De Ruysscher D, Pijls-Johannesma M, Vansteenkiste J, Kester A, Rutten I, Lambin P. Systematic review and meta-analysis of randomised, controlled trials of the timing of chest radiotherapy in patients with limited-stage, small-cell lung cancer. Ann Oncol. 2006 Apr;17(4):543-52. doi: 10.1093/annonc/mdj094. Epub 2005 Dec 12. PMID 16344277
- [Background] De Ruysscher D, Pijls-Johannesma M, Bentzen SM, Minken A, Wanders R, Lutgens L, Hochstenbag M, Boersma L, Wouters B, Lammering G, Vansteenkiste J, Lambin P. Time between the first day of chemotherapy and the last day of chest radiation is the most important predictor of survival in limited-disease small-cell lung cancer. J Clin Oncol. 2006 Mar 1;24(7):1057-63. doi: 10.1200/JCO.2005.02.9793. PMID 16505424
- [Background] Xia B, Chen GY, Cai XW, Zhao JD, Yang HJ, Fan M, Zhao KL, Fu XL. Is involved-field radiotherapy based on CT safe for patients with limited-stage small-cell lung cancer? Radiother Oncol. 2012 Feb;102(2):258-62. doi: 10.1016/j.radonc.2011.10.003. Epub 2011 Nov 5. PMID 22056536
- [Background] van Loon J, De Ruysscher D, Wanders R, Boersma L, Simons J, Oellers M, Dingemans AM, Hochstenbag M, Bootsma G, Geraedts W, Pitz C, Teule J, Rhami A, Thimister W, Snoep G, Dehing-Oberije C, Lambin P. Selective nodal irradiation on basis of (18)FDG-PET scans in limited-disease small-cell lung cancer: a prospective study. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):329-36. doi: 10.1016/j.ijrobp.2009.04.075. Epub 2009 Sep 24. PMID 19782478
- [Background] Kies MS, Mira JG, Crowley JJ, Chen TT, Pazdur R, Grozea PN, Rivkin SE, Coltman CA Jr, Ward JH, Livingston RB. Multimodal therapy for limited small-cell lung cancer: a randomized study of induction combination chemotherapy with or without thoracic radiation in complete responders; and with wide-field versus reduced-field radiation in partial responders: a Southwest Oncology Group Study. J Clin Oncol. 1987 Apr;5(4):592-600. doi: 10.1200/JCO.1987.5.4.592. PMID 3031226
- [Background] Liengswangwong V, Bonner JA, Shaw EG, Foote RL, Frytak S, Eagan RT, Jett JR, Richardson RL, Creagan ET, Su JQ. Limited-stage small-cell lung cancer: patterns of intrathoracic recurrence and the implications for thoracic radiotherapy. J Clin Oncol. 1994 Mar;12(3):496-502. doi: 10.1200/JCO.1994.12.3.496. PMID 8120547
- [Background] Miller KL, Marks LB, Sibley GS, Clough RW, Garst JL, Crawford J, Shafman TD. Routine use of approximately 60 Gy once-daily thoracic irradiation for patients with limited-stage small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):355-9. doi: 10.1016/s0360-3016(02)04493-0. PMID 12738309
- [Background] Turrisi AT 3rd, Kim K, Blum R, Sause WT, Livingston RB, Komaki R, Wagner H, Aisner S, Johnson DH. Twice-daily compared with once-daily thoracic radiotherapy in limited small-cell lung cancer treated concurrently with cisplatin and etoposide. N Engl J Med. 1999 Jan 28;340(4):265-71. doi: 10.1056/NEJM199901283400403. PMID 9920950
- [Background] Choi NC, Herndon JE 2nd, Rosenman J, Carey RW, Chung CT, Bernard S, Leone L, Seagren S, Green M. Phase I study to determine the maximum-tolerated dose of radiation in standard daily and hyperfractionated-accelerated twice-daily radiation schedules with concurrent chemotherapy for limited-stage small-cell lung cancer. J Clin Oncol. 1998 Nov;16(11):3528-36. doi: 10.1200/JCO.1998.16.11.3528. PMID 9817271
- [Background] Overgaard J, Hansen HS, Specht L, Overgaard M, Grau C, Andersen E, Bentzen J, Bastholt L, Hansen O, Johansen J, Andersen L, Evensen JF. Five compared with six fractions per week of conventional radiotherapy of squamous-cell carcinoma of head and neck: DAHANCA 6 and 7 randomised controlled trial. Lancet. 2003 Sep 20;362(9388):933-40. doi: 10.1016/s0140-6736(03)14361-9. PMID 14511925
- [Background] Bese NS, Hendry J, Jeremic B. Effects of prolongation of overall treatment time due to unplanned interruptions during radiotherapy of different tumor sites and practical methods for compensation. Int J Radiat Oncol Biol Phys. 2007 Jul 1;68(3):654-61. doi: 10.1016/j.ijrobp.2007.03.010. Epub 2007 Apr 30. PMID 17467926
- [Background] Videtic GM, Fung K, Tomiak AT, Stitt LW, Dar AR, Truong PT, Yu EW, Vincent MD, Kocha WI. Using treatment interruptions to palliate the toxicity from concurrent chemoradiation for limited small cell lung cancer decreases survival and disease control. Lung Cancer. 2001 Aug-Sep;33(2-3):249-58. doi: 10.1016/s0169-5002(00)00240-3. PMID 11551420
- [Background] Xia B, Hong LZ, Cai XW, Zhu ZF, Liu Q, Zhao KL, Fan M, Mao JF, Yang HJ, Wu KL, Fu XL. Phase 2 study of accelerated hypofractionated thoracic radiation therapy and concurrent chemotherapy in patients with limited-stage small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2015 Mar 1;91(3):517-23. doi: 10.1016/j.ijrobp.2014.09.042. Epub 2014 Dec 3. PMID 25481679
- [Background] Hou JM, Krebs MG, Lancashire L, Sloane R, Backen A, Swain RK, Priest LJ, Greystoke A, Zhou C, Morris K, Ward T, Blackhall FH, Dive C. Clinical significance and molecular characteristics of circulating tumor cells and circulating tumor microemboli in patients with small-cell lung cancer. J Clin Oncol. 2012 Feb 10;30(5):525-32. doi: 10.1200/JCO.2010.33.3716. Epub 2012 Jan 17. PMID 22253462
- [Background] Hou JM, Greystoke A, Lancashire L, Cummings J, Ward T, Board R, Amir E, Hughes S, Krebs M, Hughes A, Ranson M, Lorigan P, Dive C, Blackhall FH. Evaluation of circulating tumor cells and serological cell death biomarkers in small cell lung cancer patients undergoing chemotherapy. Am J Pathol. 2009 Aug;175(2):808-16. doi: 10.2353/ajpath.2009.090078. Epub 2009 Jul 23. PMID 19628770
- [Background] Hiltermann TJN, Pore MM, van den Berg A, Timens W, Boezen HM, Liesker JJW, Schouwink JH, Wijnands WJA, Kerner GSMA, Kruyt FAE, Tissing H, Tibbe AGJ, Terstappen LWMM, Groen HJM. Circulating tumor cells in small-cell lung cancer: a predictive and prognostic factor. Ann Oncol. 2012 Nov;23(11):2937-2942. doi: 10.1093/annonc/mds138. Epub 2012 Jun 11. PMID 22689177